CLINICAL TRIAL: NCT01908140
Title: A Randomised, Double-blind, Double-dummy, Active-controlled Study Evaluating the Efficacy, Safety and Tolerability of Twice-daily Aclidinium Bromide/Formoterol Fumarate Compared With Twice-daily Salmeterol/Fluticasone Propionate for 24 Weeks Treatment in Symptomatic Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Study of Aclidinium Bromide/Formoterol Fumarate Compared With Salmeterol/Fluticasone Propionate in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M/40464/39; 2013-000116-14 (EudraCT Number)
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Results first posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — aclidinium bromide; Formoterol Fumarate; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aclidinium Bromide / Formoterol Fumarate (Experimental): Aclidinium Bromide 400 μg / Formoterol Fumarate 12 μg BID for 24 Weeks
  Interventions: Drug: Aclidinium Bromide / Formoterol Fumarate
- Salmeterol / Fluticasone propionate (Active Comparator): Salmeterol 50 μg / Fluticasone propionate 500 μg BID for 24 Weeks
  Interventions: Drug: Salmeterol / Fluticasone

INTERVENTIONS:
Drug: Aclidinium Bromide / Formoterol Fumarate
  Arms: Aclidinium Bromide / Formoterol Fumarate
Drug: Salmeterol / Fluticasone
  Other Names: Seretide; Advair
  Arms: Salmeterol / Fluticasone propionate

SUMMARY:
The purpose of the study is to compare the efficacy, safety and tolerability of aclidinium bromide/formoterol fumarate and salmeterol/fluticasone propionate in patients with chronic obstructive pulmonary disease (COPD)

ELIGIBILITY:
Inclusion Criteria:

* Adult male or non-pregnant, non-lactating female aged ≥40.
* Current or ex-cigarette smoker, with a smoking history of at least 10 pack-years
* Patients with a clinical diagnosis of COPD according to GOLD guidelines 2013, with a post-bronchodilator FEV1 <80%, and FEV1/FVC < 70% at Screening Visits
* Symptomatic patients with a COPD assessment test (CAT) ≥10 at Screening and Randomisation Visits
* Patient must be able to perform repeatable pulmonary function testing for FEV1 according to ATS/ERS 2005 criteria at Screening Visits
* Patients eligible and able to participate in the trial and who consent to do so in writing after the purpose and nature of the investigation have been explained

Exclusion Criteria:

* History or current diagnosis of asthma
* Development of a respiratory tract infection or COPD exacerbation within 6 weeks (or 3 months if hospitalisation was required) before the Screening Visit or during the run-in period
* Clinically significant respiratory conditions
* Type I or uncontrolled Type II diabetes, uncontrolled hypo- or hyperthyroidism, hypokalaemia, or hyperadrenergic state, uncontrolled or untreated hypertension
* Patients who, in the investigator's opinion, may need to start a pulmonary rehabilitation programme during the study and/or patients who started/finished it within 3 months prior to Screening Visit
* Use of long-term oxygen therapy (≥15 hours/day)
* Patients treated on daily basis with triple therapy (LABA+LAMA+ICS) within 4 weeks prior to the Screening Visit
* Patient who does not maintain regular day/night, waking/sleeping cycles including night shift workers
* Clinically significant cardiovascular conditions
* Patient with clinically relevant abnormalities in the results of the clinical laboratory tests, ECG parameters or in the physical examination at the Screening Visit
* Patient with a history of hypersensitivity reaction to inhaled anticholinergics, sympathomimetic amines, or inhaled medication or any component thereof (including report of paradoxical bronchospasm)
* Patient with known narrow-angle glaucoma, symptomatic bladder neck obstruction, acute urinary retention, or patients with symptomatic non-stable prostatic hypertrophy
* Patient with known non-controlled history of infection with human immunodeficiency virus (HIV) and/or active hepatitis
* History of malignancy of any organ system (including lung cancer), treated or untreated, within the past 5 years other than basal or squamous cell skin cancer
* Patient with any other serious or uncontrolled physical or mental dysfunction
* Patient with a history (within 2 years prior to Screening Visit) of drug and/or alcohol abuse that may prevent study compliance based on investigator judgment
* Patient unlikely to be cooperative or that can't comply with the study procedures
* Patient treated with any investigational drug within 30 days (or 6 half-lives, whichever is longer) prior to Screening Visit
* Patient who intend to use any concomitant medication not permitted by this protocol or who have not undergone the required stabilization periods for prohibited medication
* Any other conditions that, in the investigator's opinion, might indicate the patient to be unsuitable for the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 933 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Garcia, Ph.D., Study Director — Global Medicines Development
Locations (108):
- Austria (5):
  - Almirall Investigational Site, Feldbach
  - Almirall Investigational Site, Feldkirch
  - Almirall Investigational Site, Grieskirchen
  - Almirall Investigational Site, Linz
  - Almirall Investigational Site, Salzburg
- Bulgaria (8):
  - Almirall Investigational Site, Dimitrovgrad
  - Almirall Investigational Site, Gabrovo
  - Almirall Investigational Site, Kozloduy
  - Almirall Investigational Site, Petrich
  - Almirall Investigational Site, Plovdiv
  - Almirall Investigational Site, Razgrad
  - Almirall Investigational Site, Stara Zagora
  - Almirall Investigational Site, Vidin
- Canada (6):
  - Almirall Investigational Site, Edmonton, Alberta
  - Almirall Investigational Site, Vancouver, British Columbia
  - Almirall Investigational Site, Moncton, New Brunswick
  - Almirall Investigational Site, Toronto, Ontario
  - Almirall Investigational Site, Saint Romuald, Quebec
  - Almirall Investigational Site, Trois-Rivières, Quebec
- Czechia (6):
  - Almirall Investigational Site, Karlovy Vary
  - Almirall Investigational Site, Kralupy nad Vltavou
  - Almirall Investigational Site, Liberec
  - Almirall Investigational Site, Ostrava - Hrabuvka
  - Almirall Investigational Site, Rokycany
  - Almirall Investigational Site, Strakonice
- France (3):
  - Almirall Investigational Site, Nîmes
  - Almirall Investigational Site, Perpignan
  - Almirall Investigational Site, Vieux-Condé
- Germany (21):
  - Almirall Investigational Site, Berlin
  - Almirall Investigational Site, Bochum
  - Almirall Investigational Site, Bonn
  - Almirall Investigational Site, Cologne
  - Almirall Investigational Site, Cottbus
  - Almirall Investigational Site, Dortmund
  - Almirall Investigational Site, Dresden
  - Almirall Investigational Site, Frankfurt
  - Almirall Investigational Site, Gauting
  - Almirall Investigational Site, Großhansdorf
  - Almirall Investigational Site, Hamburg
  - Almirall Investigational Site, Hanover
  - Almirall Investigational Site, Jena
  - Almirall Investigational Site, Leipzig
  - Almirall Investigational Site, Marburg
  - Almirall Investigational Site, Munich
  - Almirall Investigational Site, Rüdersdorf
  - Almirall Investigational Site, Schwabach
  - Almirall Investigational Site, Wiesbaden
  - Almirall Investigational Site, Wiesloch
  - Almirall Investigational Site, Witten
- Hungary (9):
  - Almirall Investigational Site, Balassagyarmat
  - Almirall Investigational Site, Budapest
  - Almirall Investigational Site, Debrecen
  - Almirall Investigational Site, Komárom
  - Almirall Investigational Site, Nyíregyháza
  - Almirall Investigational Site, Pécs
  - Almirall Investigational Site, Százhalombatta
  - Almirall Investigational Site, Szigetszentmiklós
  - Almirall Investigational Site, Vásárosnamény
- Italy (3):
  - Almirall Investigational Site, Pisa
  - Almirall Investigational Site, Pordenone
  - Almirall Investigational Site, Trieste
- Lithuania (3):
  - Almirall Investigational Site, Kaunas
  - Almirall Investigational Site, Klaipėda
  - Almirall Investigational Site, Vilnius
- Netherlands (6):
  - Almirall Investigational Site, Almere Stad
  - Almirall Investigational Site, Beek
  - Almirall Investigational Site, Eindhoven
  - Almirall Investigational Site, Hoofddorp
  - Almirall Investigational Site, Leeuwarden
  - Almirall Investigational Site, Rotterdam
- Poland (15):
  - Almirall Investigational Site, Bialystok
  - Almirall Investigational Site, Gdansk
  - Almirall Investigational Site, Katowice
  - Almirall Investigational Site, Krakow
  - Almirall Investigational Site, Lodz
  - Almirall Investigational Site, Ostrowiec Świętokrzyski
  - Almirall Investigational Site, Piła
  - Almirall Investigational Site, Poznan
  - Almirall Investigational Site, Proszowice
  - Almirall Investigational Site, Sopot
  - Almirall Investigational Site, Szczecin
  - Almirall Investigational Site, Tarnów
  - Almirall Investigational Site, Tczew
  - Almirall Investigational Site, Warsaw
  - Almirall Investigational Site, Wilkowice-Bystra
- South Africa (6):
  - Almirall Investigational Site, Belville
  - Almirall Investigational Site, Cape Town
  - Almirall Investigational Site, Gauteng
  - Almirall Investigational Site, Middelburg
  - Almirall Investigational Site, Pretoria
  - Almirall Investigational Site, Somerset West
- Spain (9):
  - Almirall Investigational Site, Alicante
  - Almirall Investigational Site, Barcelona
  - Almirall Investigational Site, Elda
  - Almirall Investigational Site, Laredo
  - Almirall Investigational Site, Madrid
  - Almirall Investigational Site, Palma de Mallorca
  - Almirall Investigational Site, Sant Boi de Llobregat
  - Almirall Investigational Site, Santander
  - Almirall Investigational Site, Seville
- United Kingdom (8):
  - Almirall Investigational Site, Birmingham
  - Almirall Investigational Site, Chorley
  - Almirall Investigational Site, Glasgow
  - Almirall Investigational Site, Liverpool
  - Almirall Investigational Site, Manchester
  - Almirall Investigational Site, Middlesex
  - Almirall Investigational Site, Reading
  - Almirall Investigational Site, Sidcup

REFERENCES:
- [Derived] Vogelmeier C, Paggiaro PL, Dorca J, Sliwinski P, Mallet M, Kirsten AM, Beier J, Seoane B, Segarra RM, Leselbaum A. Efficacy and safety of aclidinium/formoterol versus salmeterol/fluticasone: a phase 3 COPD study. Eur Respir J. 2016 Oct;48(4):1030-1039. doi: 10.1183/13993003.00216-2016. Epub 2016 Aug 4. PMID 27492833
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3947&filename=LAC39_CSR_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 140 activated sites. A total of 121 sites randomised patients. The first patient was screened in Oct 2013 and the last patient visit was in Aug 2014.
Pre-assignment Details: Patients fulfilling inclusion/exclusion criteria at the time of the screening visit were entered into a run-in period of 14-21 days to assess disease stability.
Groups:
- Aclidinium Bromide / Formoterol Fumarate: Experimental: Aclidinium Bromide / Formoterol Fumarate Aclidinium Bromide 400 μg / Formoterol Fumarate 12 μg BID for 24 Weeks
- Salmeterol / Fluticasone: Active Comparator: Salmeterol / Fluticasone propionate Salmeterol 50 μg / Fluticasone propionate 500 μg BID for 24 Weeks
Period: Overall Study
Arm/Group | Aclidinium Bromide / Formoterol Fumarate | Salmeterol / Fluticasone
Started | 468 | 465
Completed | 402 | 386
Not Completed | 66 | 79
Not completed — Other or Progressive Disease | 5 | 12
Not completed — Lack of Efficacy | 7 | 5
Not completed — Withdrawal by Subject | 23 | 24
Not completed — Lost to Follow-up | 1 | 6
Not completed — Protocol Violation | 8 | 9
Not completed — Adverse Event | 22 | 23

BASELINE CHARACTERISTICS:
Population: Patients with more than 1 treatment were analysed in the Safety population with the actual treatment assigned; for this reason, the Overall Number of Baseline Participants in the safety population is different than the randomised population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aclidinium Bromide / Formoterol Fumarate | Salmeterol / Fluticasone | Total
Number analyzed (Participants) | 467 | 466 | 933
Age, Customized [Mean (Standard Deviation); unit: years]
  Age (years), mean (SD) | 63.5 (8.1) | 63.3 (7.5) | 63.4 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 166 | 326
  Male | 307 | 300 | 607
Region of Enrollment [Number; unit: participants]
  Austria | 23 | 24 | 47
  Bulgaria | 30 | 32 | 62
  Canada | 12 | 6 | 18
  Czech Republic | 11 | 14 | 25
  France | 10 | 4 | 14
  Germany | 118 | 136 | 254
  Hungary | 50 | 48 | 98
  Italy | 6 | 5 | 11
  Lithuania | 17 | 10 | 27
  Netherlands | 11 | 11 | 22
  Poland | 67 | 55 | 122
  South Africa | 68 | 66 | 134
  Spain | 28 | 34 | 62
  United Kingdom | 16 | 21 | 37

OUTCOME MEASURES:

1. Primary Outcome: Peak Forced Expiratory Volume in One Second (FEV1) at Week 24
Description: Peak FEV1 define at the highest value observed in the 3h after the morning IMP administration
Time Frame: At Week 24
Population: ITT population: randomized patients who took at least one dose of IMP and have a baseline FEV1 assessment.
  PP population: subset of ITT constituted by patients who met all inclusion/exclusion criteria liable to affect the efficacy ssessment, attained sufficient compliance to treatment and did not present serious deviations of the protocol.
Measure: Least Squares Mean (Standard Error); unit: Liters
Units Other Than Participants: participants
Arm/Group | Aclidinium Bromide / Formoterol Fumarate | Salmeterol / Fluticasone
Number analyzed (Participants) | 389 | 376
Liters | 1.655 (0.011) | 1.562 (0.011)
Statistical Analysis 1: Comparison: Aclidinium Bromide / Formoterol Fumarate vs Salmeterol / Fluticasone; This sample size of 900 had 90% power to show that the lower bound of the two-sided 95% confidence interval for the difference between Aclidinium bromide 400 μg/Formoterol Fumarate 12 μg and SeretideTM AccuhalerTM (50/500 μg) in Peak FEV1 at 24 weeks is above -0,055 L; Test type: Non-Inferiority or Equivalence — non-inferiority margin=-0,055 L; p < 0.001, MMRM; If non-inferiority on the PP was achieved then switch to superiority was tested on the ITT; Mean Difference (Final Values) = 0.093, 95% CI 2-sided [0.063 to 0.123]

2. Secondary Outcome: Transition Dyspnoea Index (TDI) Focal Score at Week 24
Description: The TDI includes the same 3 categories as BDI and 7 ratings indicating the magnitude of the change from baseline in each category: from -3 ("major deterioration") to zero ("no change") to +3 ("major improvement"). Category scores are added to compute the Focal Score (from -9 to 9)
Time Frame: At Week 24
Population: PP population defined as a subset of ITT constituted by patients who met all inclusion/exclusion criteria liable to affect the efficacy ssessment, attained sufficient compliance to treatment and did not present serious deviations of the protocol.
Measure: Least Squares Mean (Standard Error); unit: TDI Focal Score
Units Other Than Participants: participants
Arm/Group | Aclidinium Bromide / Formoterol Fumarate | Salmeterol / Fluticasone
Number analyzed (Participants) | 353 | 341
TDI Focal Score | 1.9 (0.17) | 1.9 (0.17)
Statistical Analysis 1: Comparison: Aclidinium Bromide / Formoterol Fumarate vs Salmeterol / Fluticasone; The total sample size provided 81% nominal power to show that the lower bound of the two-sided 95 confidence interval for the difference between Aclidinium bromide 400 μg/Formoterol fumarate 12 μg and SeretideTM AccuhalerTM (50/500 μg) in transitional dyspnoea index (TDI) at 24 weeks is above -0,5; Test type: Non-Inferiority or Equivalence — non-inferiority limit -0.5 units; p > 0.05, MMRM; Mean Difference (Final Values) = -0.001, 95% CI 2-sided [-0.46 to 0.46]

ADVERSE EVENTS:
Time Frame: 24 Weeks treatment + 2 weeks follow-up (±3 days)
Arm/Group | Aclidinium Bromide / Formoterol Fumarate | Salmeterol / Fluticasone
Serious Adverse Events (participants affected / at risk) | 35/467 | 33/466
Other Adverse Events (participants affected / at risk) | 124/467 | 135/466
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aclidinium Bromide / Formoterol Fumarate (N=467) | Salmeterol / Fluticasone (N=466)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cor Pulmonale (Cardiac disorders) | 1 (1) | 0 (0)
Artrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Artrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmogenic right ventricular dysp (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Endometritis (Infections and infestations) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 4 (4)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract and infection (Infections and infestations) | 0 (0) | 1 (1)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Grastroenteritis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Squamous cell carcinoma of head (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Schizoaffective disorder depressive (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Adnexa uteri mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
COPD (exacerbation) (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 8 (9)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Subclavian artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aclidinium Bromide / Formoterol Fumarate (N=467) | Salmeterol / Fluticasone (N=466)
Nasopharyngitis (Infections and infestations) | 26 (30) | 28 (33)
Headache (Nervous system disorders) | 28 (42) | 32 (46)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 70 (82) | 75 (81)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the information related to this clinical trial is considered strictly confidential and is the property of AstraZeneca. This information will not be given to a third party without the written consent of AstraZeneca. Publication and/or presentation, whether complete or partial, of any part of the data or results of this trial will be subject to revision and written agreement between the investigator and AstraZeneca.